CLINICAL TRIAL: NCT06354283
Title: The Effect of Progressive Muscle Relaxation Exercises Applied to Women With Low Sexual Satisfaction on Sexual Satisfaction and Functioning of Women and Their Partners: A Randomized Controlled Trial
Brief Title: Progressive Muscle Relaxation Exercises Women With Low Sexual Satisfaction Sexual Satisfaction and Functioning of Women and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Progresif
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Women With Low Sexual Satisfaction; Partners of Women With Low Sexual Satisfaction
Keywords: Sexual Satisfaction; Progressive Muscle Relaxation Exercises; Sexual Functioning
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Intervention Model Description: Intervention Group and Control Group
Who Masked: Investigator, Outcomes Assessor
Masking Description: The progressive relaxation intervention and follow-up was conducted by the researcher who was not blinded to the interventions (PSI). Randomization was performed by another academic who was not an investigator in the study. In order to avoid bias, the researcher who conducted the intervention did not participate in any step of the pre-test, post-test and statistical evaluation process. Group information was not shared with the statistician who performed the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Progressive muscle relaxation techniques were explained to the women from the couples assigned to the Intervention Group by a researcher. In addition to relaxation exercises, deep breathing movements were also explained to the women and progressive muscle relaxation exercises and breathing exercises were performed together. The importance of the exercises and how to do them were explained to the women for about 30 minutes by the researcher and then demonstrated practically for 30 minutes. Each progressive muscle relaxation exercise session lasted approximately 20-25 minutes. The women in the intervention group continued the exercises at home three times a week for four weeks. The women in the intervention group were telephoned once a week by the researcher to provide reminders and counseling regarding the study
  Interventions: Behavioral: Progressive Muscle Relaxation Exercises
- Control (No Intervention): The study was announced on social media and online to identify women and men who met the sample selection criteria. Couples who scored between 20-40 on the New Sexual Satisfaction Scale for women and 11 or higher on the Arizona Sexual Life Scale for men and women were randomized into two groups. A data collection form was applied to the couples included in the sample.
  The Control Group was followed up by continuing the daily routine. At the end of two and four weeks, the New Sexual Satisfaction Scale and Arizona Sexual Life Scale were administered to all women and their partners.

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation Exercises — Progressive muscle relaxation techniques were explained to the women from the couples assigned to the Intervention Group by a researcher. In addition to relaxation exercises, deep breathing movements were also explained to the women and progressive muscle relaxation exercises and breathing exercises were performed together. The importance of the exercises and how to do them were explained to the women by the researcher for about 30 minutes and then demonstrated practically for 30 minutes. Each progressive muscle relaxation exercise session lasted approximately 20-25 minutes. The women in the intervention group continued the exercises at home three times a week for four weeks.
  Arms: Intervention

SUMMARY:
This study was conducted to investigate the effect of progressive muscle relaxation exercises on sexual satisfaction and functioning of women and their partners in women with low sexual satisfaction.

Method: The single-blind, randomized controlled study was conducted between April 2023 and January 2024. The sample of the study was women with low sexual satisfaction and their partners were randomized into two groups as intervention and control. Each group consisted of 120 couples, n=60. The women in the intervention group were given progressive muscle relaxation techniques three times a week for four weeks. The results of the study focused on the effect on sexual satisfaction and functioning of men and women.

DETAILED DESCRIPTION:
This study was conducted to investigate the effect of progressive muscle relaxation exercises on sexual satisfaction and functioning of women and their partners in women with low sexual satisfaction.

Hypotheses H1: Progressive muscle relaxation techniques increase sexual satisfaction in women with low sexual satisfaction.

H2: Progressive muscle relaxation techniques positively affect sexual function in women with low sexual satisfaction.

H3: Progressive muscle relaxation techniques increase sexual satisfaction of partners in women with low sexual satisfaction.

H4: Progressive muscle relaxation techniques positively affect sexual function of partners in women with low sexual satisfaction.

While the population of the study consisted of women aged 18-35 years, the minimum sample size was calculated using G Power. Accordingly, it was found that the number of women to be sampled should be 44 for each group, totaling 88 women. Considering that there would be losses, the sample was planned to be 60 couples for each group, totaling 120 couples. There were no losses during the study.

Sample Selection Criteria; Women who had an active sexual life, were of childbearing age (18-35 years), had the same partner for the last year, had not given birth before, and scored between 20-40 on the New Sexual Satisfaction Scale were included.

Sample Exclusion Criteria; Women and their partners who had chronic gynecological diseases, whose own and/or partner used psychiatric drugs, who were pregnant during the study, who had diagnoses that prevented sexuality such as vaginusmus, erectile dysfunction, etc., who scored below 11 on the Arizona Sexual Life Scale were not included in the study.

The study was announced on social media and online to identify women and men who met the sample selection criteria. Couples who scored between 20-40 on the New Sexual Satisfaction Scale for women and 11 or higher on the Arizona Sexual Life Scale for men and women were randomized into two groups. A data collection form was applied to the couples included in the sample.

Progressive muscle relaxation techniques were explained to the women from the couples assigned to the Intervention Group by a researcher. In addition to relaxation exercises, deep breathing movements were also explained to the women and progressive muscle relaxation exercises and breathing exercises were performed together. The importance of the exercises and how to do them were explained to the women by the researcher for about 30 minutes and then demonstrated practically for 30 minutes. Each progressive muscle relaxation exercise session lasted approximately 20-25 minutes. The women in the intervention group continued the exercises at home three times a week for four weeks. The women in the intervention group were telephoned once a week by the researcher to provide reminders and counseling about the study (Progressive muscle relaxation steps were given as an additional file).

The Control Group was followed up by continuing the daily routine. At the end of two and four weeks, the New Sexual Satisfaction Scale and Arizona Sexual Life Scale were administered to all women and their partners.

ELIGIBILITY:
Inclusion Criteria:

* Women who had active sexual life, were of childbearing age (18-35 years), had the same partner for the last year, had not given birth before, and scored between 20-40 on the New Sexual Satisfaction Scale were included.

Exclusion Criteria:

* Women and their partners who had chronic gynecological diseases, who were using psychiatric medication for themselves and/or their partners, who were pregnant at the time of the study, who had diagnoses that hindered sexuality such as vaginismus, erectile dysfunction, etc., and who scored below 11 on the Arizona Sexual Life Scale were not included in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women and their partners with low sexual satisfaction
Enrollment: 120 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Sexual Satisfaction | Pre-intervention, 2nd and 4th weeks after intervention
  The scale consists of 20 items. The 5-point Likert-type scale is scored as (1) I am not satisfied at all (2) I am somewhat satisfied (3) I am moderately satisfied (4) I am very satisfied (5) I am extremely satisfied. The lowest score that can be obtained from the scale is 20 and the highest score is 100. The scale consists of a self-centered sub-dimension and a partner/ sexual activity-centered sub-dimension. These two subscales represent the New Sexual Satisfaction Scale. The self-centered sub-dimension consists of items 1-10 and the partner/ sexual activity-centered sub-dimension consists of items 11-20. Scoring is calculated by summing the items. A high score on the scale indicates good sexual satisfaction. There are no reverse scored items in the scale.

SECONDARY OUTCOMES:
Sexual Function | Pre-intervention, 2nd and 4th weeks after intervention
  It was used to include women and men in the sample and to evaluate sexual function during follow-up. The scale, which has separate male and female forms, is filled in by the patients and no special training is required for its interpretation. The scale consists of five items on a six-point Likert scale with a score range of 5-30 and an increase in the total score indicates sexual dysfunction. According to Soykan, a scale score of ≥11 is the cut-off point for sexual dysfunction. In the validity and reliability study in Turkey, the scale was found to have high internal consistency and reliability with Cronbach's α values of 0.89-0.90 and to be valid in differentiating sexual dysfunction. In this study, it was 0.78 in men and 0.82 in women.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Şule Bilgiç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is appropriate to present it after publication